CLINICAL TRIAL: NCT07009223
Title: Lifestyle Interventions to Prevent cOgnitive Deficits in Subjects With Depressive Symptoms: From mEchanisms to Clinical pRactice
Acronym: POWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); University of Milan (Other); China Medical University, China (Other); University College Cork (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CERP-2024-23685718
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder (MDD); Physical Activity; Inflammation; Metabolome; Gut Microbiota; Depressive Symptoms
Keywords: Depression; Cognition; nutrition
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity; Inflammation; Depression | interventions — Diet, Mediterranean; Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Control group (CON) (Active Comparator)
  Interventions: Behavioral: Mediterranean Diet
- Group 2: CON + physical activity (Experimental)
  Interventions: Behavioral: Mediterranean Diet; Behavioral: Physical Activity
- Group 3: CON + Cognitive training (Experimental)
  Interventions: Behavioral: Mediterranean Diet; Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Mediterranean Diet — Participants will receive only the educational intervention about the Mediterranean diet. The program consists of 4-5 online sessions conducted by a nutritionist.
Behavioral: Physical Activity — In addition to educational sessions on the Mediterranean diet, there will be 2-3 weekly personalized exercise sessions, followed by a dedicated personal trainer at a partner gym. The treatment will last 12 weeks.
  Arms: Group 2: CON + physical activity
Behavioral: Cognitive Training — In addition to educational sessions on the Mediterranean diet, there will be one weekly cognitive training session in groups, supervised by qualified staff at the IRCCS FBF. The treatment will last for 12 weeks.
  Arms: Group 3: CON + Cognitive training

SUMMARY:
The goal of this clinical study is to investigate if lifestyle changes can help prevent cognitive decline and reduce depressive symptoms in people between the ages of 50 and 80 with depressive symptoms or a diagnosis of major depression, but without signs of cognitive decline.

The main questions it aims to answer are:

* Does regular physical activity improve mood and memory in people who are depressed or have depressive symptoms?
* Does cognitive training help prevent mental difficulties in people at risk of cognitive decline?
* Do changes in diet and lifestyle alter the composition of the gut microbiota and immuno-related infiammatory factors?

Researchers will compare three different treatment groups to see which intervention is most effective in improving mental and cognitive health.

The participants:

* Will take part to online sessions on healthy eating based on the Mediterranean diet
* Some will do regular exercise, supervised by a personal trainer
* Others will do weekly cognitive training in small groups at the hospital
* They will provide blood and fecal samples and complete cognitive tests and clinical questionnaires at the beginning, at the end of the treatment (12 weeks), and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 80 years;
* Diagnosis of DDM according to DSM-5 or depressive symptoms (PHQ-9 or GDS-15 ≥ 5, the choice of test will be justified by the participant's age);
* Ability to provide written informed consent.

Exclusion Criteria:

* Active gastrointestinal disorders;
* Autoimmune disorders;
* Chronic inflammatory disorders;
* Diagnosis of dementia; cognitive impairment or mild functional impairment.
* Use of antibiotics and/or anti-inflammatory drugs in the 8 weeks prior to the screening visit.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
MADR Scale for Depression | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-administered scale designed to assess the severity of depressive symptoms. It consists of 10 items, each rated on a scale from 0 to 6, yielding a total score ranging from 0 to 60. Higher scores indicate greater severity of depression, meaning a worse clinical outcome.
PHQ-9 | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered instrument used to assess the severity of depressive symptoms based on DSM criteria. It consists of 9 items, each rated from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 27. Higher scores reflect more severe depressive symptoms, indicating a worse clinical outcome.
GDS-15 | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Geriatric Depression Scale - Short Form (GDS-15) is a self-report questionnaire designed to screen for depressive symptoms in older adults. It contains 15 yes/no items, with a total score ranging from 0 to 15. Higher scores indicate more severe depressive symptoms, representing a worse clinical outcome.
WHOQOL-BREF | Baseline, Week 12, and 3-month follow-up (Week 24)
  The World Health Organization Quality of Life - Bref (WHOQOL-BREF) is a self-report questionnaire developed by the WHO to assess quality of life across multiple domains. It contains 26 items rated on a 5-point Likert scale. Higher scores indicate a better quality of life, reflecting a more favorable outcome.
RBANS | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Repeatable Battery for the Assessment of Neuropsychological (RBANS) is a neuropsychological battery composed of 12 subtests grouped into five domains: Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory. It yields index scores and a total scale score. Higher scores indicate better cognitive functioning, reflecting a more favorable clinical outcome.
TMT | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Trail Making Test (TMT) evaluates processing speed (Part A) and executive function, including task switching (Part B). The outcome is the time (in seconds) required to complete each part. Lower completion times indicate better performance and cognitive flexibility.
DSST | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Digit Symbol Substitution Test (DSST) evaluates attention, processing speed, and working memory. Participants match numbers and symbols in a limited time. Higher scores reflect better performance.
M-WCST | Baseline, Week 12, and 3-month follow-up (Week 24)
  The Modified Wisconsin Card Sorting (M-WCST) measures cognitive flexibility and executive function. Outcomes include number of categories completed and perseverative errors. More categories and fewer errors indicate better performance.

SECONDARY OUTCOMES:
Immunitary-related factors levels | Baseline, Week 12, and 3-month follow-up (Week 24)
  Plasma/serum levels of cytokines
Gut Microbiome Composition | Baseline, Week 12, and 3-month follow-up (Week 24)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy